CLINICAL TRIAL: NCT01161641
Title: " An Open Label Pilot Study Evaluating Safety and Evidence of Therapeutic Effect of IV Admin of 2-0, 3-0 Desulfated Heparin, Treatment of Exacerbation of Protein Losing Enteropathy (PLE) Associated With Single Ventricle Palliative Surgery"
Brief Title: Pilot/Ph I Safety and Efficacy of ODSH in Protein Losing Enteropathy Secondary to Single Ventricle Palliative Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Extremely slow accural due to rarity of medical condition studied.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGX-ODSH-2009-PLE
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2015-08

CONDITIONS: Protein Losing Enteropathy
Keywords: Protein Losing Enteropathy
MeSH Terms: conditions — Protein-Losing Enteropathies | interventions — KPNA1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ODSH at 0.125 mg/kg/h (Experimental): First cohort of 3 subjects to be administered the lowest dose of ODSH.
  Interventions: Drug: ODSH at 0.125 mg/kg/h
- ODSH at 0.250 mg/kg/h (Experimental): Second cohort of 3 subjects to receive the medium dose of ODSH
  Interventions: Drug: ODSH at 0.250 mg/kg/h
- ODSH at 0.375 mg/kg/h (Experimental): Third and last cohort of subject to receive the high dose of ODSH.
  Interventions: Drug: ODSH at 0.375 mg/kg/h

INTERVENTIONS:
Drug: ODSH at 0.125 mg/kg/h — ODSH 1000 mg vials containing 20 cc of normal saline (50 mg/ml) to be prepared for 96-h IV infusion with normal saline based on subject's weight and dose assigned by Study Cohort 1 of 0.125 mg/kg/h.
  Other Names: Cohort 1
  Arms: ODSH at 0.125 mg/kg/h
Drug: ODSH at 0.375 mg/kg/h — ODSH 1000 mg vials containing 20 cc of normal saline (50 mg/ml) to be prepared for 96-h IV infusion with normal saline based on subject's weight and dose assigned by Study Cohort 3 of 0.375 mg/kg/h.
  Other Names: Cohort 3
  Arms: ODSH at 0.375 mg/kg/h
Drug: ODSH at 0.250 mg/kg/h — ODSH 1000 mg vials containing 20 cc of normal saline (50 mg/ml) to be prepared for 96-h IV infusion with normal saline based on subject's weight and dose assigned by Study Cohort 2 of 0.250 mg/kg/h.
  Other Names: Cohort 2
  Arms: ODSH at 0.250 mg/kg/h

SUMMARY:
Protein Losing Enteropathy (PLE) is a serious medical condition that may develop in children and adults with congenital heart disease for which a palliative procedure known as the "Fontan procedure" has been performed. The loss of serum proteins into the gastrointestinal tract that is associated with PLE can cause serious symptoms and life-threatening complications. A number of clinical studies have suggested that heparin administration can have clinical benefit in children with PLE, however the risk of bleeding associated with the administration of heparin is an important concern and commonly limits its administration. ODSH is a desulfated heparin with minimal anticoagulation properties but which, in pre-clinical studies, appears to have the potential to replace heparin and greatly reduce the risk of bleeding. This open label study is to assess the safety and evidence of therapeutic effect of the administration of ODSH as a 4-day continuous intravenous infusion in patients with an exacerbation of their PLE.

DETAILED DESCRIPTION:
Protein Losing Enteropathy (PLE)is a serious and sometimes fatal condition that develops in approximately 10% of children who have undergone the single ventricle palliative surgery known as the Fontan procedure. The mechanisms by which PLE develops are not fully understood, however a recent mechanism has been proposed consistent with the specific loss of heparan sulfate proteoglycans from the basolateral surface of the intestinal epithelial cells resulting in the loss of serum protein including albumin and immunoglobulins into the gastrointestinal tract that is associated with protein losing enteropathy. A number of clinical studies have suggested that heparin administration can have clinical benefit in children with PLE, however the risk of bleeding as a consequence of treatment is an important concern and commonly limits its administration. ODSH (2-0, 3-0 desulfated heparin) is a modified heparin that preserves the anti-inflammatory properties of heparin with minimal or no anticoagulation effects. ODSH has been studied in the rodent model of PLE an has shown improvement of PLE in this model due to restoration of heparan sulfate and Syndecan 1 with stabilization of the cell matrix of the capillary endothelium.

This open label clinical study will enroll 9 subjects with a dose escalation (3 doses) study design. Three subjects will be treated with the lower dose of ODSH then an ad hoc safety committee will assess the safety information to make a recommendation regarding advancing to the next higher dose of ODSH until, if appropriate, the 3 dose cohorts have been completed. Plasma albumin and fecal alpha 1 antitrypsin which are both biological markers of protein loss through the intestinal lumen in this condition, are the primary variables that will be evaluated as evidence of a therapeutic effect together with the improvement of PLE signs and symptoms. The effect of ODSH on the associated diarrhea, abdominal pain, and peripheral edema or ascites will be evaluated using visual/categorical scales for the patients to assess symptoms and clinical evaluation by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 6 years old.
2. History of single ventricle palliative surgery.
3. Anticipated need for four or more days of hospitalization, in the investigator's judgment, for the treatment of exacerbation of PLE.

   Clinically significant PLE is defined as the presence of clinically significant symptoms (including, but not limited to, diarrhea, abdominal pain, peripheral edema and/or ascites), AND increased fecal alpha 1-antitrypsin (FA1AT; > 200 mg/dl) OR hypoalbuminemia of < 3 gr/dL; requiring supplemental albumin infusions.
4. Prothrombin time (PT) and activated partial thromboplastin time (aPTT) not higher than 1.25 times the ULN for age.
5. Platelet count of > 80,000 per mm3, hemoglobin of > 9.5 g/dL.
6. The adult subject or the underage subject/legal guardian is willing to provide informed consent and to comply with the study procedures.
7. Female subject of childbearing potential who is not pregnant, and is not lactating and is not planning to become pregnant during the study and will use medically acceptable contraception method for the duration of the study.

Exclusion Criteria:

1. Has congenital or acquired hematologic disease or coagulation disorder.
2. Has other type of PLE not associated with single ventricle palliative surgery e.g. subjects with congenital defects of glycation or with Crohn's disease; congenital trypsinogen or enterokinase deficiency;
3. Has a clinical need for prophylactic or therapeutic treatment with oral or parenteral anticoagulant medications within 72 hours from the start of ODSH treatment or during the study. [The use of antithrombotic agents such as acetyl salicylic acid for cardiovascular prophylaxis or clopidogrel (or similar drug class agents) is permitted].
4. Has documented liver failure or a serum ALT or AST greater than 1.5 times the upper limit of normal, or total bilirubin greater than 1.5 the upper limit of normal;
5. Has clinically significant proteinuria or severe renal failure based on a creatinine clearance < 30 mL/min calculated from plasma creatinine (Appendix B) with the Cockcroft-Gault formula for adults or with any of the recommended formulas for subjects 6 to 18 years old;
6. Has active gastrointestinal ulcer disease or evidence of gastrointestinal bleeding or urinary tract bleeding or any other source of bleeding within 60 days of the Screening visit.
7. History of HIV, hepatitis B or hepatitis C; and
8. Major surgery, stroke or myocardial infarction within the past 60 days from screening. Subjects with recent minor surgery can be enrolled in the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of PLE symptoms and signs. | Day 4 after 96 hours of IV continuous infusion of ODSH
  Clinical Improvement of signs & symptoms of PLE such as diarrhea, abdominal pain, peripheral edema, and ascites. Visual/categorical scales will be used by the study subjects and the investigators to assess diarrhea/abdominal pain intensity as well as The Global Impression of Improvement. The investigator will assess peripheral edema and ascites.
Fecal alpha 1 antitrypsin (FA1AT) | Day 4 after 96 hours of ODSH IV continuous infusion
  Decrease of Fecal alpha 1 antitrypsin level at Day 4 compared to baseline.
Serum albumin levels. | Day 4 after 96 hours of continuous IV infusion of ODSH
  Serum albumin levels at Day 4 compared to Baseline. A serum albumin level of 3 or more mg/dL or at least an increase of 25% from baseline at Day 4 or the reduction in the need for additional albumin infusions will be considered as clinically significant.
ODSH safety | Day 1, 2, 3 and 4
  aPTT as a measure of coagulation effect from ODSH will be measured every day. If the aPTT value is 8 or more seconds higher than the upper limit of normal value of aPTT for the study site then the ODSH infusion rate will be decreased as recommended in the protocol. Coagulation and bleeding abnormalities will be monitored closely by the investigator. Liver enzymes will also be monitored during the study.

SECONDARY OUTCOMES:
PK: ODSH plasma blood levels at steady state | Day 3 (during Day 3 of ODSH IV continuous infusion)
  Assess the plasma levels of ODSH at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Mark Russell, MD, Principal Investigator — Division of Pediatric Cardiology, University of Michigan Health System
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles ( Gastroenterology & Nutrition), Los Angeles, California
  - Department of Cardiology, Children's Hospital Boston, Boston, Massachusetts
  - Division of Pediatric Cardiology, University of Michigan Health System, Ann Arbor, Michigan
  - Sanford Children's ( Sanford Research / USD), Sioux Falls, South Dakota